CLINICAL TRIAL: NCT02973295
Title: Silymarin® - Efficacy in Treatment of Non-alcoholic Fatty Liver Disease (NAFLD) Controlled by Laboratory and and Elastographic Parameters
Brief Title: Silymarin in NAFLD
Acronym: SINF
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Sponsor withdrawn their agreement
Sponsor: University Hospital Rijeka (Other)
Collaborators: University of Rijeka, Medical Faculty (Unknown); Belupo (Other); University of Rijeka, Faculty of Health studies (Unknown)
Responsible Party: Principal Investigator, Goran Hauser, Goran Hauser, Principal investigator, University Hospital Rijeka
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KBCRi/2016-GH01
Record Dates: First submitted 2016-11-04; First posted 2016-11-25 (Estimated); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Non-Alcoholic Fatty Liver Disease
Keywords: NAFLD;; Fibroscan; Silymarin
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease | interventions — Silymarin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Silymarin (Experimental): Silymarin 2x200 mg 8 weeks (2x2 caps) Silymarin 2x100 mg 16 weeks (2x1 caps)
  Interventions: Drug: Silymarin
- Group Placebo (Placebo Comparator): 2x2 placebo caps 8 weeks 2x1 placebo caps 16 weeks
  Interventions: Other: Placebo Oral Capsule

INTERVENTIONS:
Drug: Silymarin — Capsules contains 100 mg of silymarin
  Arms: Group Silymarin
Other: Placebo Oral Capsule — Capsule will be identical in shape, size and color, packed in the same way like verum
  Other Names: no other names
  Arms: Group Placebo

SUMMARY:
This study evaluates the influence of Silymarin in reducing laboratory, ultrasonographic (Fibroscan) and metabolic components of NAFLD. Half of the patients will receive Silymarin (Verum) while the other half will receive placebo

DETAILED DESCRIPTION:
In this study will participate patients who come to the regular ambulatory examinations (referred by gastroenterologists, nephrologists or family physicians in the Department of Gastroenterology and Department of Nephrology, dialysis and kidney transplantation KBC Rijeka) and have one or more components of the metabolic syndrome (hypertension, diabetes, obesity, dyslipidemia).Nonalcoholic fatty liver disease will be defined by transient elastography (FibroScan, Echosens, Paris); Controlled Attenuation Parameter (CAP) for assesment of liver steatosis and Liver Stiffness Measurements (LSM) for liver fibrosis. In all patients other causes of chronic liver disease will be excluded; chronic viral hepatitis, autoimmune diseases and other metabolic liver diseases as well as use of drugs than can cause liver steatosis and fibrosis and alcoholic liver disease.

This study will include 350 patients. Taking into account the possible drop-out rate around 15% of the patients during the study period, a total of 400 patients will be randomized. Patients will be randomized into two groups. The first group will be consisted of the patients with NAFLD who will be receiving Verum therapy during the 6 month period. The second group will be consisted of the patients with NAFLD who will be receiving placebo during the 6 months period, which will be identical to the Verum preparation in its packaging and form.

After the 6 months of therapy in all patients will be evaluated: liver enzymes and metabolic laboratory parameters of NAFLD (insulin resistance, lipidogram and serum glucose), as well as the TE-CAP in order to evaluate the efficiency of Silymarin for the treatment of NAFLD.

ELIGIBILITY:
Inclusion Criteria:

* NAFLD patients
* signed informed consent
* possibility to follow instruction and the protocol

Exclusion Criteria:

* chronic B or C hepatitis
* usage of hepatotoxic drugs in the period of 6 months before inclusion
* chronic kidney insufficiency (grade 4 and 5), hemodialysis
* any other chronic liver disease
* opioid dependancy
* any malignancy
* HIV seropositivity
* alcohol abuse
* pregnancy
* inability to follow the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-12 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Change (Reduction) of parameters of liver steatosis defined by CAP (Controlled Attenuation Parameter) and liver fibrosis defined by LSM (liver stiffness measurements) during the 6 months period | 0 week (Initiation) and during 24-25 week (End of the Study)
  Transient elastography detected by FibroScan®, Echosense, France

SECONDARY OUTCOMES:
Change in liver enzymes in period of 6 months | 0 week (Initiation) and during 24-25 week (End of the Study)
  AST (Aspartate Aminotransferase ) ALT (alanine aminotransferase), GGT (gamma-glutamyltransferase), ALP (Alkaline Phosphatase). All outcomes have the same units of measure (UI/L) and all together represents liver function test.
Change in insulin resistance in period of 6 months | 0 week (Initiation) and during 24-25 week (End of the Study)
  In the assessment of the insulin resistance HOMA-IR scoring system will be used (fasting insulin (microU/L) x fasting glucose (nmol/L)/22.5.)
Change in lipidogram in period of 6 months | 0 week (Initiation) and during 24-25 week (End of the Study)
  lipidogram (total cholesterol, LDL-cholesterol, HDL-cholesterol and triglycerides) All outcomes have the same units of measure (umol/L) and all together represents lipid profile

CONTACTS AND LOCATIONS:
Overall Officials: Goran Hauser, MD, PhD, Principal Investigator — Clinical Hospital Centre Rijek, Croatia
Locations (1):
- Clinical Hospital Centre, Rijeka, Kresimirova 42, Croatia

IPD SHARING:
Plan to Share IPD: Yes
All patient data will be available to other researchers after interim analysis

REFERENCES:
- [Background] Festi D, Schiumerini R, Marzi L, Di Biase AR, Mandolesi D, Montrone L, Scaioli E, Bonato G, Marchesini-Reggiani G, Colecchia A. Review article: the diagnosis of non-alcoholic fatty liver disease -- availability and accuracy of non-invasive methods. Aliment Pharmacol Ther. 2013 Feb;37(4):392-400. doi: 10.1111/apt.12186. Epub 2012 Dec 20. PMID 23278163
- [Background] Mikolasevic I, Orlic L, Franjic N, Hauser G, Stimac D, Milic S. Transient elastography (FibroScan((R))) with controlled attenuation parameter in the assessment of liver steatosis and fibrosis in patients with nonalcoholic fatty liver disease - Where do we stand? World J Gastroenterol. 2016 Aug 28;22(32):7236-51. doi: 10.3748/wjg.v22.i32.7236. PMID 27621571
- [Background] Mikolasevic I, Milic S, Orlic L, Stimac D, Franjic N, Targher G. Factors associated with significant liver steatosis and fibrosis as assessed by transient elastography in patients with one or more components of the metabolic syndrome. J Diabetes Complications. 2016 Sep-Oct;30(7):1347-53. doi: 10.1016/j.jdiacomp.2016.05.014. Epub 2016 May 20. PMID 27324703
- [Background] Mikolasevic I, Orlic L, Hrstic I, Milic S. Metabolic syndrome and non-alcoholic fatty liver disease after liver or kidney transplantation. Hepatol Res. 2016 Aug;46(9):841-52. doi: 10.1111/hepr.12642. Epub 2016 Feb 4. PMID 26713425